CLINICAL TRIAL: NCT00925561
Title: Predictors of Coronary Artery Calcification in an African American Cohort
Brief Title: Examining the Genetic Predictors of Coronary Artery Calcification in African Americans
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of Mississippi Medical Center (Other); Wake Forest University (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Patricia Peyser, Professor of Epidemiology, University of Michigan
Other Study IDs: 643; R01HL085571 (NIH); 5R01HL085571 (NIH)
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Atherosclerosis
Keywords: Coronary Artery Calcification
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood to measure risk factors and stored DNA for genetic studies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
Coronary artery disease (CAD) is an important health concern for African Americans, who are diagnosed with CAD at high rates. Coronary artery calcification, which is characterized by calcium deposits in the coronary arteries, is a contributing factor to CAD. This study will examine the possible genetic causes of coronary artery calcification in African Americans.

DETAILED DESCRIPTION:
In the United States, more people die from CAD than any other disease, with African Americans, particularly women and young men, being more affected by CAD than European Americans. One cause of CAD is atherosclerosis, a condition in which deposits of fat, cholesterol, and other substances build up along the inner walls of arteries. Coronary artery calcification occurs as a result of atherosclerosis and is characterized by calcium build up in the arteries. Non-invasive imaging, including computed tomography (CT) scans, of coronary artery calcification is an effective way to assess CAD risk. The Genetic Epidemiology Network of Arteriopathy (GENOA) study, which is part of the Family Blood Pressure Program (FBPP), is a study that examined siblings with high blood pressure during two exams conducted between 1995 and 2004. The purpose of this new GENOA study, which will enroll past GENOA participants, is to identify genetic factors that may lead to the development of coronary artery calcification in African Americans. Conducting genetic studies in the African American population will result in greater understanding of the mechanisms of atherosclerosis, and may lead to improved strategies for the early identification of people at risk for CAD and the development of new treatments for CAD.

This study will enroll people who have participated in the second GENOA exam and who live in Jackson, Mississippi. Participants will attend one study visit at the University of Mississippi Medical Center. During the study visit, participants will be interviewed by study staff about their medical and family health history; health behaviors; physical activity levels; and use of tobacco, alcohol, and medications. They will complete a walking activity and tasks to assess memory, thinking speed, and accuracy. Participants will also complete a questionnaire about their mood, a physical examination, a CT scan of the heart, and a blood collection. A portion of blood will be stored for future research studies.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the second GENOA exam in Jackson, Mississippi and is alive and willing to participate

Exclusion Criteria:

* Reported a history of heart attack, stroke, or coronary or non-coronary heart surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will come from Jackson, MS and will include all men and women belonging to sibships that previously participated in the second GENOA exam. The sampling frame includes 1482 African Americans in 627 sibships providing 1552 sibling pairs from Jackson, Mississippi.
Sampling Method: Non-Probability Sample
Enrollment: 752 (Actual)
Dates: Start 2009-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Coronary Artery Calcification | Measured during participants' single study visit

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Peyser, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States